CLINICAL TRIAL: NCT02020538
Title: Does Varying the Chloride Content of Intravenous Fluid Alter the Risk of Acute Kidney Injury After Cardiac Surgery?
Brief Title: Limiting IV Chloride to Reduce AKI After Cardiac Surgery
Acronym: LICRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Australian and New Zealand College of Anaesthetists (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 382/13
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2019-12

CONDITIONS: Patients Undergoing Cardiothoracic Surgery
Keywords: Thoracic surgery; cardiac surgery; acute kidney injury; hyperchloremia; intravenous fluid
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, prospective, open-label, 4-period sequential study
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloride-rich IV fluid (Placebo Comparator): The chloride-rich strategy will include 0.9% saline as the perioperative crystalloid of choice with 4% albumin as the perioperative colloid of choice.
  Interventions: Other: High-chloride perioperative intravenous fluid strategy
- Chloride-poor IV fluid (Active Comparator): A low-chloride strategy of perioperative IV fluid will include PlasmaLyte 148 or Hartmann's solution as the crystalloid of choice with 20% albumin as the colloid of choice.
  Interventions: Other: Low-chloride perioperative intravenous fluid strategy

INTERVENTIONS:
Other: Low-chloride perioperative intravenous fluid strategy — The low-chloride perioperative IV fluid strategy will include the use of PlasmaLyte 148 or Hartmann's solution as the crystalloid of choice and 20% albumin as the colloid of choice.
  Other Names: Chloride-poor IV fluid
  Arms: Chloride-poor IV fluid
Other: High-chloride perioperative intravenous fluid strategy
  Other Names: Chloride-rich IV fluid
  Arms: Chloride-rich IV fluid

SUMMARY:
This primary aim of this study is to test the impact of a strategy of perioperative chloride-restriction through intravenous (IV) fluid therapy on the incidence of acute kidney injury after cardiac surgery.

A prospective, open-label, single-centre 4-period sequential study of varying strategies of perioperative IV fluid composition will test the hypothesis that a perioperative protocol for the administration of chloride-poor intravenous fluids compared to chloride-rich intravenous fluids will reduce the incidence of AKI after adult cardiothoracic surgery.

DETAILED DESCRIPTION:
After an initial run-in period of approximately 1 month (using a chloride-rich fluid strategy), the first study period of 5 months will commence, also comprising a chloride-rich perioperative IV fluid therapy strategy (0.9% saline or 4% albumin). This will include intraoperative fluid and postoperative fluid for the duration of stay in the intensive care unit. This will then be followed by a 1-month transition period before a second period of 5 months will commence where perioperative intravenous fluid therapy will consist of chloride-poor fluids (Lactated Ringer's solution or concentrated 20% albumin). A subsequent 1-month transition period will then be followed by a third period of 5 months characterized by perioperative IV fluid therapy with an alternative combination of chloride-poor solutions (PlasmaLyte® 148 or concentrated 20% albumin). A final 1-month transition period will be followed by a fourth and final period of 5 months characterized by a return to perioperative IV fluid therapy with chloride-rich fluids (0.9% saline or 4% albumin). A final 1-month run-off period using a chloride-rich perioperative fluid strategy will follow prior to study completion.

ELIGIBILITY:
Inclusion Criteria:

All adult patients undergoing surgery by Division of cardiothoracic surgery

Exclusion Criteria:

Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1298 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2015-12-09 (Actual); Study Completion 2016-02-12 (Actual)

PRIMARY OUTCOMES:
Peak ∆ serum creatinine | 5 days postoperatively
  Maximum change in serum creatinine from baseline
AKI ≥stage2 | 5 days postoperatively
  AKI, ≥stage2, defined by creatinine-based KDIGO criteria

SECONDARY OUTCOMES:
Individual stages of AKI | 7 days
  Individual stages of AKI, defined by creatinine-based KDIGO criteria
Mortality | On discharge from hospital (7-30 days)
  Mortality
Renal replacement therapy | On discharge from hospital (7-30 days)
  Renal replacement therapy
ICU Length of stay | On discharge from hospital (7-30 days)
  ICU Length of stay
Hospital Length of stay | On discharge from hospital (7-30 days)
  Hospital Length of stay
Time to first extubation | On discharge from hospital (7-30 days)
  Time to first extubation
Red cell transfusion requirement | Intraoperative and postoperatively through completion of postoperative day 1 or ICU discharge, whichever occurred first
  Volume of packed red blood cells transfused
Fresh frozen plasma transfusion requirement | Intraoperative and postoperatively through completion of postoperative day 1 or ICU discharge, whichever occurred first
  Volume of fresh frozen plasma transfused
Platelet transfusion requirement | Intraoperative and postoperatively through completion of postoperative day 1 or ICU discharge, whichever occurred first
  Volume of platelets transfused
Cryoprecipitate transfusion requirement | Intraoperative and postoperatively through completion of postoperative day 1 or ICU discharge, whichever occurred first
  Volume of cryoprecipitate transfused

OTHER OUTCOMES:
Time-weighted mean serum chloride concentration | First 5 days and through ICU admission
  A time-weighted calculation of mean serum chloride concentration
Incidence of hypernatremia | On discharge from hospital (7-30 days)
  Incidence of hypernatremia (SNa+ >150 mmol/L)
Incidence of hyponatremia | On discharge from hospital (7-30 days)
  Incidence of hyponatremia (SNa+ <130 mmol/L)
Incidence of hyperchloremia | On discharge from hospital (7-30 days)
  Incidence of hyperchloremia (SCl- >110 mmol/L)
Incidence of hypochloremia | On discharge from hospital (7-30 days)
  Incidence of hypochloremia (SCl- <96 mmol/L)
Incidence of acidemia | On discharge from hospital (7-30 days)
  Incidence of acidemia (pH <7.3)
Incidence of alkalemia | On discharge from hospital (7-30 days)
  Incidence of alkalemia (pH >7.5)

CONTACTS AND LOCATIONS:
Overall Officials: David R McIlroy, MBBS, MClinEpi, FANZCA, Principal Investigator — Alfred Hospital and Monash University
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] McIlroy DR, Murphy D, Shotwell MS, Bhatia D. Peak Serum Chloride and Hyperchloremia in Patients Undergoing Cardiac Surgery Is Not Explained by Chloride-Rich Intravenous Fluid Alone: A Post-Hoc Analysis of the LICRA Trial. J Cardiothorac Vasc Anesth. 2021 May;35(5):1321-1331. doi: 10.1053/j.jvca.2020.07.085. Epub 2020 Aug 7. PMID 32863142
- [Derived] McIlroy D, Murphy D, Kasza J, Bhatia D, Wutzlhofer L, Marasco S. Effects of restricting perioperative use of intravenous chloride on kidney injury in patients undergoing cardiac surgery: the LICRA pragmatic controlled clinical trial. Intensive Care Med. 2017 Jun;43(6):795-806. doi: 10.1007/s00134-017-4772-6. Epub 2017 Mar 25. PMID 28343236